CLINICAL TRIAL: NCT00247286
Title: A Randomised, Single-Blind Comparison of Pelvic Floor Muscle Exercises With Biofeedback Versus Weighted Vaginal Cones in the Management of Genuine Stress Incontinence : A Pilot Study
Brief Title: Weighted Vaginal Cones Versus Biofeedback in the Treatment of Urodynamic Stress Incontinence: a Randomized Trial.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Marie-Andree Harvey, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OBGY-076-00
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Incontinence, Stress
Keywords: urodynamic stress incontinence; weighted vaginal cones; pelvic floor biofeedback; randomized controlled trial
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- a (Experimental): Weighted vaginal cones used to perform pelvic floor exercises
  Interventions: Behavioral: weighted vaginal cones
- b (Active Comparator): Biofeedback
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Behavioral: weighted vaginal cones
  Arms: a
Behavioral: Biofeedback — Pelvic floor muscles exercises performed with a biofeedback machine
  Arms: b

SUMMARY:
The purpose of this study is to determine the objective (urodynamic) cure rates and effect on patient quality of life after six months of treatment for two different nonsurgical management options for genuine stress urinary incontinence in females: weighted vaginal cones and formal supervised pelvic floor physiotherapy with biofeedback.

Hypothesis: Assuming a minimum of six months of treatment, weighted vaginal cones are as effective as a formal supervised program of pelvic floor physiotherapy with biofeedback for the treatment of uncomplicated genuine stress urinary incontinence in females.

DETAILED DESCRIPTION:
Background and Rationale Urinary incontinence is a widespread and debilitating medical problem, with an estimated prevalence of between 17-45% in adult women. Genuine stress incontinence is the most common form of urinary incontinence in women, with objective diagnosis made via urodynamics. Urinary continence is maintained when the urethral resistance (pressure) is greater than the intravesical pressure. Genuine stress incontinence occurs when pressure transmission to the urethra is compromised by poor anatomic support of the proximal urethra resulting from weakened pelvic floor musculature and/or defective endopelvic fascia. While the gold standard for treatment of genuine stress incontinence is still considered to be surgical, there is renewed interest among both patients and surgeons for nonsurgical (conservative) management. The goal of conservative therapy is to restrengthen and retrain the pelvic floor muscles to improve urethral pressure transmission and thus improve the continence mechanism.

Nonsurgical therapies include PFME with or without biofeedback, and weighted vaginal cones. PFME with biofeedback are widely accepted as an effective conservative treatment for genuine stress incontinence, with subjective cure rates estimated to be as high as 70 percent. However, to date, objective cure rates as defined by urodynamics have not been well documented. Similarly, while limited studies suggest that vaginal cone therapy results in a subjective cure rate of 60%, objective cure rates still have not been determined. With growing clinic and surgical waiting lists and rising hospital costs, weighted vaginal cones, if objectively proven to be a comparably effective alternative to physiotherapy, will offer an effective management option for stress incontinence, thus, perhaps avoiding referral to a tertiary hospital for physiotherapy, and surgery.

We hypothesize that following a minimum of six months of treatment, weighted vaginal cones would be as effective as a formal supervised program of pelvic floor physiotherapy with biofeedback for the treatment of uncomplicated genuine stress urinary incontinence in females. We are thus seeking to evaluate the feasibility of a randomized clinical trial.

Method

An estimated 60 women identified from ambulatory clinics with multichannel urodynamics documenting genuine stress urinary incontinence will be needed to participate in this single-blind, randomized pilot study. Once entered, patients will be randomized to receive one of two different nonsurgical treatments: PFME with biofeedback or weighted vaginal cones. The patients will chart compliance to treatment for the duration of the study. A quality of life questionnaire will be completed at the beginning and end of the trial, along with a subjective assessment of incontinence severity via a standardized questionnaire. The study period will be six months. Upon completion of the study, patients will undergo repeat multichannel urodynamics and perineal pad testing to determine if genuine stress incontinence is present or absent and thus whether objective cure has been achieved. Results will be analyzed and compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* Females, between the ages of 18-65 years, will be entered into this study. Additional inclusion criteria are a history of urinary stress incontinence and multichannel cystometry confirming the presence of genuine stress incontinence (GSI).

Exclusion Criteria:

* urodynamic identification detrusor instability
* active (untreated or resistant) urinary tract infection
* any other disease that is felt by the investigators to potentially interfere with participation (e.g. arthritis limiting dexterity and thus interfering with the insertion and removal of vaginal cones)
* previous treatment with pelvic floor physiotherapy with biofeedback or functional electric stimulation for urinary incontinence
* previous use of weighted vaginal cones
* previous anti-incontinence surgery
* significant pelvic organ prolapse or those with abnormal vaginal anatomy (the Pelvic Organ Prolapse Quantification (POP-Q) system of scoring for prolapse will be used, Grade > III)
* use of concomitant treatments during the trial or the start of new medications that may alter continence mechanism
* inability to understand instructions in French or English or provide informed consent (e.g., psychiatric disease).
* pregnancy (which may alter pelvic anatomy may over the course of the study and thus make evaluation of treatment methods impossible)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2001-09; Primary Completion 2007-01 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Urodynamic studies | 6 months

SECONDARY OUTCOMES:
Cough stress test | 6 months
Standardized fixed bladder volume pad test | 6 months
I-QOL questionnaire | 6 months
Urogenital Distress Inventory | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Andree Harvey, MD MSc, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided